CLINICAL TRIAL: NCT06555601
Title: A First-in-Human, Randomized, Investigator-Blind, Participant-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of UCB3101 in Healthy Participants
Brief Title: A First-in-human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of UCB3101 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: safety reasons
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: UP0124; 2023-504586-24 (Registry Identifier: EU Clinical Trials); U1111-1305-5063 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-07-25; First posted 2024-08-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: UCB3101

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 1) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 2 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 2) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 3 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 3) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 4 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 4) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 5 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 5) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 6 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 6) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 7 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 7) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo
- Cohort 8 (Experimental): Study participants randomized to this arm will receive a single dose of UCB3101 (Dose 8) or placebo.
  Interventions: Drug: UCB3101; Drug: Placebo

INTERVENTIONS:
Drug: UCB3101 — Study participants will receive UCB3101 as prespecified in each cohort.
Drug: Placebo — Study participants will receive placebo as prespecified in each cohort to maintain the blinding.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a single ascending dose of UCB3101 in cohorts of healthy male and female study participants.

ELIGIBILITY:
* Participants must be 18 to 65 years of age inclusive, at the time of signing the informed consent form (ICF).
* Participants are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
* Participants with clinical laboratory test results within the reference ranges of the laboratory. Isolated test results that are outside the specified ranges and that are deemed clinically nonsignificant are allowed at the discretion of the investigator (except for liver enzymes). If a participant has 1 isolated test result outside the specific range for which the clinical significance is uncertain, repeat testing may be allowed at the discretion of the investigator.
* Participants are non-tobacco users or have given up smoking for at least 6 months prior to Screening.
* Participants have received a COVID-19 vaccine, including 2 boosters.
* Participants with body weight within 50.0 to 110.0kg and body mass index within the range 18.0 to 30.0kg/m2 (~40 to 66lbs/m2) (inclusive).
* Participant is male or female.

  1. Male participants must refrain from donating sperm for the duration of the study and for 3 months after planned completion of the study. A male participant with a female partner who is a woman of childbearing potential (WOCBP) must agree to use contraception for the duration of the study and for 3 months after planned completion of the study.
  2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and either not a WOCBP or a WOCBP who agrees to follow the contraceptive guidance for the duration of the study and for 1 month after planned completion of the study.
* Participant must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF.
* Participant must be considered reliable and capable of adhering to the protocol, according to the judgment of the investigator, and capable of communicating satisfactorily with the investigator and complying with all study requirements.

Exclusion Criteria:

* Vulnerable individuals (eg, individuals kept in detention, serving soldiers), employees of the Sponsor or the contract research organization (CRO), with direct involvement in the proposed study or other studies under the direction of the investigator or the CRO, as well as family members of the employees or the investigator
* Participant has any medical or psychiatric condition that jeopardize or would compromise the study participant's ability to participate in this study.
* Participant has any clinically significant Electrocardiogram (ECG) abnormalities.
* Participant has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months.
* History or presence of clinically significant respiratory, neurological, gastrointestinal, renal, hepatic, pancreatic, hematological, cardiovascular, musculoskeletal, genitourinary, immunological, or dermatological disorders.
* Participant has had prior history of lymphoma, leukemia, or any malignancy.
* Participant has a clinically significant active infection (eg, sepsis, pneumonia, abscess) or has had a serious infection within 4 weeks before the first dose of IMP.
* Participant has had recurrent (at least 2) clinically relevant infections (eg, tooth abscess, opportunistic infections, boils, etc) in the past 6 months.
* Participant has a history of recurrent headaches, including migraine.
* Participant has evidence or history of significant active bleeding or coagulation disorder.
* Participant has a history of chronic alcohol or drug abuse within 12 months prior to Baseline.
* Participant has a history of skin disorders or extensive tattooing that prevent clear visibility of the skin in case of a hypersensitivity reaction.
* Participant has scheduled surgery between Screening and 1 month after end of study visit.
* Participant has a history of clinically significant back pain, back pathology, and/or back injury that may predispose participant to complications or technical difficulty with lumbar puncture (LP).
* Participant has medical or surgical conditions for which LP is contraindicated.
* Participant is allergic to lidocaine or its derivatives.
* Participant has any clinically relevant brain magnetic resonance imaging (MRI) abnormality at Screening.
* Participant has received any prescription or nonprescription medicines, including any monoclonal antibody (mAb) therapies and over the counter remedies or herbal and dietary supplements (other than vitamins within recommended daily dose limits) within 14 days (or 5 half-lives of the respective drug, whichever is longer) prior to Baseline, other than occasional use of analgesics such as paracetamol or topical nasal corticosteroids for seasonal rhinitis.
* Participant has participated in another study of an investigational medicinal product (IMP) within 90 days (or 5 half-lives of the drug, whichever is longer) prior to Baseline or is currently participating in another study of an IMP.
* Participant has prior exposure to any IMP specifically targeting triggering receptor expressed on myeloid cells 1 (TREM1).
* Participant has received any live vaccination within the 8 weeks prior to Day 1 or is anticipated to do so within 120 days after the final dose of IMP.
* Participant has any clinically relevant abnormal findings in physical examination, laboratory tests, vital signs, or ECG.
* Participant has total bilirubin >upper limit of normal (ULN).
* Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Participant has a positive urine test for substances of abuse.
* Participant has a known active mycobacterium tuberculosis (TB) disease.
* Participant has a known history of active TB involving any organ system unless adequately treated.
* Participant has a positive laboratory test results for human immunodeficiency virus-1/2 antibodies), hepatitis B surface antigen, or hepatitis B core antibody result at Screening.
* Participant has a positive hepatitis C antibody test result at Screening or within 3 months prior to Baseline.
* Participant has clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Participant has symptomatic herpes zoster within 3 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of any treatment- emergent adverse events (TEAE) | From Baseline to Safety Follow-up (up to Week 21)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Incidence of any treatment-emergent Serious Adverse Events (SAE) | From Baseline to Safety Follow-up (up to Week 21)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death;
  * Is life-threatening; Requires inpatient hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect;
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients or may require medical or surgical intervention to prevent any of the above.
Incidence of discontinuation from treatment due to treatment- emergent adverse events (TEAE) | From Baseline to Safety Follow-up (up to Week 21)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Maximum Serum Concentration (Cmax) of UCB3101 | From Day 1 (Predose) up to Week 21
  Maximum serum concentration (Cmax) of UCB3101 will be reported.
Area Under the Serum Concentration-Time Curve (AUC) of UCB3101 | From Day 1 (Predose) up to Week 21
  Area under the serum concentration-time curve (AUC) of UCB3101 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- UP0124 1, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual participant-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.